CLINICAL TRIAL: NCT04518124
Title: Neoadjuvant Trial on the Efficacy of Propranolol Monotherapy in Cutaneous Angiosarcoma
Brief Title: Propranolol in Angiosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Anticancer Fund, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N19PCA
Record Dates: First submitted 2020-06-09; First posted 2020-08-19 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Angiosarcoma
Keywords: Propranolol; Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propranolol (Experimental)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol will be administered as monotherapy in a dose of 40-80 mg 2-3 times a day, if tolerated. The study consists of a single arm.

SUMMARY:
This is a window opportunity study of propranolol in patients with angiosarcoma. The aim of this study is to prospectively evaluate the activity of propranolol in the clinical setting as monotherapy, where the neoadjuvant setting provides a good opportunity to rapidly evaluate both the clinical response and histological response, without a significant delay in anti-cancer treatment.

DETAILED DESCRIPTION:
A pilot neoadjuvant window of opportunity study will be performed to explore the activity of propranolol monotherapy in angiosarcoma. The study consists of a single arm. Propranolol will be administred as monotherapy in a dose of 40-80 mg 2-3 times a day, if tolerated. When patients are diagnosed, standard anti-cancer treatment will be scheduled in 6 weeks while propranolol treatment can start immediately after diagnosis and will be continued until the day the standard anti-cancer treatment is started. The duration of treatment will therefore be 3-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of angiosarcoma
2. Patients with primary, recurrent and metastasised disease are eligible;
3. Patients with a window of at least 3 weeks before surgery or systemic therapy;
4. Age ≥ 18 years;
5. Able and willing to give written informed consent;
6. WHO performance status of 0, 1 or 2;
7. Evaluable disease according to RECIST 1.1 criteria; radiologic visible disease is not obligated in patients with cutaneous angiosarcoma
8. Minimal acceptable safety laboratory values
9. ANC of ≥ 1.5 x 109 /L
10. Platelet count of ≥ 100 x 109 /L
11. Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ASAT and ALAT ≤ 2.5 x ULN
12. Renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (by Cockcroft-Gault formula);
13. At least one tumor lesion accessible to safely biopsy per clinical judgement of the treating physician

Exclusion Criteria:

1. Contraindication for propranolol therapy, like severe hypotension or bradycardia, sicksinus syndrome, second or third grade heart block, cardiogenic shock, untreated heart failure, severe peripheral vascular disease asthma or other obstructive lung diseases, untreated pheochromocytoma, metabolic acidosis, prolonged fasting.
2. Current treatment with β-blockade therapy.
3. Any anticancer treatment within 30 days prior to receiving the first dose of investigational treatment; with the exception of hormonal therapy for breast cancer.
4. Concurrent treatment with an anticancer therapy: with the exception of hormonal therapy for breast cancer.
5. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the investigator would impair study compliance;
6. Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications;
7. Pregnancy;
8. Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Clinical response | From start to end of treatment: 3-6 weeks
  A response is defined as CR, PR, or SD with an improvement in clinical characteristics

SECONDARY OUTCOMES:
Histological response on propranolol treatment | through study completion, an average of 2 years
  The histologic response defined as a decrease of >30% of Ki-67 index between pre- and post-propranolol treatment biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Winan van Houdt, MD PhD, Principal Investigator — Netherlands Cancer Institute - Antoni van Leeuwenhoek; Neeltje Steeghs, MD PhD, Principal Investigator — Netherlands Cancer Institute - Antoni van Leeuwenhoek
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands